CLINICAL TRIAL: NCT01345825
Title: A Randomized Controlled Trial: The Effectiveness of 8-weeks Progressive Strength Training to Patients With Unicompartmental Knee Replacement, Initiated Within the First Postoperative Week
Brief Title: Early Progressive Strength Training to Patients With Unicompartmental Knee Replacement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M-20100185
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthrosis; unicompartmental knee replacement; knee; resistance training; Muscle power; gait analysis; gait; physiotherapy; Gyro sensor
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- resistance training (Experimental)
  Interventions: Other: Resistance training

INTERVENTIONS:
Other: Resistance training — Week 1: 2 sets x 12 repetitions at 12 RM Week 2: 3 sets of 12 repetitions with 12 RM Week 3: 3 sets of 10 repetitions with 10 RM Week 4-5: 3 sets of 10 repetitions with 10 RM Week 6: 3 sets of 8 repetitions with 8 RM Week 7: 4 sets of 8 repetitions with 8 RM Week 8: 4 sets of 8 repetitions with 8 RM

SUMMARY:
The purpose and Study hypotheses:

The purpose of the study is to investigate the effect of progressive resistance training in the early postoperative phase on patients who has had unicompartmental knee replacement. The hypotheses are that this group compared to a control group will achieve greater muscle strength and functional ability in terms of gait and working capacity.

Study design:

The subjects will be randomized into two groups; intervention and control. Intervention group: strength training two times a week supervised by a physiotherapist.

Control group: Training at home, following extradited guidelines.

Endpoint:

Primary endpoint is two months postoperative. The following test will be used: muscle power test (by a Power Rig), instrumented gait analysis using a combined accelerometer and gyro-sensor in; 6 min. walk test, stair climbing test, 20 meter walking test and block step test.

Furthermore, the questionnaire KOOS will be used for monitoring every 2 weeks.

Sample size:

The power calculation is based on an expected improvement in muscle power by 25%. The risk of a type 1 error is set to 5 %, and the power is set to 80%. The calculations showed that 24 patients are needed in both groups, but 30 patient will be included in both groups to account for dropouts.

Perspectives:

This study is, to our knowledge, the first study to investigate the effect of strength training after unicompartmental knee replacement. Moreover it has , to our knowledge not been. At the moment no guidelines for rehabilitation exist, and research showed that this group of patients has a decreased function in their daily living compared with the background population. If, as expected, cases have an overall increased function compared to controls, this study can provide a basis for future rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* medial osteoarthrosis in knee assigned to unicompartmental knee replacement
* 18+ years.

Exclusion Criteria:

* rheumatoid arthritis
* neuro muscular conditions
* alcohol or drug abuse
* cognitive problems
* patients not fluid in the Danish language
* walking disability caused by other than in condition in question

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2011-03; Primary Completion 2013-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Muscle power test (by a power rig) | prior to operation (baseline), 9 weeks post operativ and 1 year post operative

SECONDARY OUTCOMES:
Gait quality | prior to operation (baseline), 9 weeks post operativ and 1 year post operative
  Instrumentet gait analysis using a combined gyro-sensor and accelerometer - inertia measurement unit(IMU).

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Søballe, Principal Investigator — Orthopaedic Surgery Research Unit, Aarhus
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark